CLINICAL TRIAL: NCT06356584
Title: Fruquintinib Combined With Sintilimab ± Radiotherapy for Third-line Treatment of Colorectal Cancer With Liver Metastases: A Randomized, Controlled, Multicenter Phase II Trial
Brief Title: Fruquintinib Combined With Sintilimab ± Radiotherapy for Third-line Treatment of Colorectal Cancer With Liver Metastases
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Shandong Cancer Hospital and Institute (Other)
Responsible Party: Principal Investigator, Jinbo Yue, Shandong Cancer Hospital Ethics Committee, Shandong Cancer Hospital and Institute
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDZLEC2024-078-01
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-01

CONDITIONS: Colorectal Cancer; Immunotherapy; Radiotherapy; Targeted Therapy; Liver Metastasis
Keywords: Colorectal cancer; Immunotherapy; Radiotherapy; Targeted therapy; Liver metastasis
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Immunotherapy; sintilimab; HMPL-013; Radiotherapy; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Immunotherapy, targert therapy, and radiotherapy (Experimental): For liver oligometastases, high-dose stereotactic body radiation therapy (SBRT) irradiation will be administered to all lesions with a dose fractionation pattern of 40-50 Gy/5F, 60-70 Gy/10F, or 65 Gy/13F. For multiple liver metastases, SBRT plus low-dose radiation therapy (LDRT) will be performed to all lesions. One or more suitable lesions (which will be selected by the physician based on proximity to organs at risk) will undergo SBRT with a dose fractionation pattern of 40-50 Gy/5F, 60-70 Gy/10F, or 65 Gy/13F, and the remaining lesions will undergo LDRT at a total dose of 1-10 Gy at 0.5-2.0 Gy/F. Extrahepatic lesions will be not treated with radiotherapy. Targeted therapy and immunotherapy will be administered one week after the end of radiation therapy. A 21-day treatment cycle of sintilimab (200 mg, D1, once every 3 weeks) will be given intravenously on day 1 of each cycle, and fruquintinib will be given on days 1 to 14.
  Interventions: Drug: Immunotherapy (Sintilimab); Drug: Targeted Therapy Agent (Fruquintinib); Radiation: Radiotherapy (SBRT and LDRT)
- Immunotherapy and targert therapy (Active Comparator): A 21-day treatment cycle of sintilimab (200 mg, D1, once every 3 weeks) will be given intravenously on day 1 of each cycle, and fruquintinib will be given on days 1 to 14.
  Interventions: Drug: Immunotherapy (Sintilimab); Drug: Targeted Therapy Agent (Fruquintinib)
- Targert therapy (Active Comparator): Treatment with fruquintinib (5 mg, po, D1-21, once every 4 weeks) will be given on days 1 through 21 in a 28-day treatment cycle.
  Interventions: Drug: Targeted Therapy Agent (Fruquintinib)

INTERVENTIONS:
Drug: Immunotherapy (Sintilimab) — Sintilimab
  Arms: Immunotherapy and targert therapy; Immunotherapy, targert therapy, and radiotherapy
Drug: Targeted Therapy Agent (Fruquintinib) — Fruquintinib
Radiation: Radiotherapy (SBRT and LDRT) — SBRT and LDRT
  Arms: Immunotherapy, targert therapy, and radiotherapy

SUMMARY:
Colorectal cancer (CRC) is a significant cause of morbidity and mortality worldwide. Its early clinical manifestations are often subtle, leading to late-stage diagnosis in about 30% of cases with distant metastases. Liver metastases are widespread and associated with poor prognosis, especially in terms of response to immunotherapy. This prospective study will evaluate the efficacy of combined therapy involving sintilimab, fruquintinib, and radiotherapy in CRC with liver metastases. The primary objectives are to assess progression-free survival, overall survival, and treatment response rates. This study aims to provide valuable insights into optimizing third-line and subsequent therapies for CRC with liver metastases by elucidating the efficacy and safety of this combined treatment approach.

DETAILED DESCRIPTION:
CRC is a significant cause of morbidity and mortality worldwide. Its early clinical manifestations are often subtle, leading to late-stage diagnosis in about 30% of cases with distant metastases. Liver metastases are widespread and associated with poor prognosis, especially in terms of response to immunotherapy. This prospective study will evaluate the efficacy of combined therapy involving sintilimab, fruquintinib, and radiotherapy in CRC with liver metastases. The primary objectives are to assess progression-free survival, overall survival, and treatment response rates. The rationale for this study stems from the intricate interplay between immunotherapy, targeted therapy, and radiotherapy in CRC management. Previous data suggest a negative correlation between liver metastases and immunotherapy efficacy, necessitating a comprehensive approach integrating multiple treatment modalities. Radiotherapy, particularly stereotactic body radiation therapy, has shown promise in controlling liver tumors and modulating the tumor microenvironment, potentially enhancing immunotherapy responses. This study aims to provide valuable insights into optimizing third-line and subsequent therapies for CRC with liver metastases by elucidating the efficacy and safety of this combined treatment approach.

ELIGIBILITY:
Inclusion Criteria:

* ECOG PS 0-2
* Histologically confirmed colorectal adenocarcinoma with liver metastases (8th edition AJCC)
* MSS/pMMR subtype
* Previously received standard first- and second-line systemic anti-tumor therapy
* At least one measurable lesion as defined by RECIST 1.1 criteria
* Access to tumor samples for biomarker assessment
* Expected survival of ≥3 months
* Normal function of major organ systems (within 14 days before enrollment)
* No systemic corticosteroid treatment within 7 days before treatment initiation, excluding physiological corticosteroid replacement therapy.
* Fertile males or females with the potential for pregnancy must use highly effective contraception methods during the trial.

Exclusion Criteria:

* Patients diagnosed with malignancies other than colorectal cancer within 3 years prior to enrollment.
* Participating in an interventional clinical study or receiving other investigational drugs or treatments with study devices within the past 4 weeks before enrollment.
* Previously received the following therapies: anti-PD-1, anti-PD-L1, or anti-PD-L2 drugs, or drugs targeting another T cell co-stimulatory or co-inhibitory receptor (e.g., CTLA-4, OX-40, CD137), fruquintinib, etc.
* Received traditional Chinese medicine or immune-modulating drugs with anti-tumor indications within the past 2 weeks before enrollment (excluding local use for controlling pleural effusion).
* Experienced active autoimmune diseases requiring systemic therapy within the past 2 years before enrollment. Replacement therapy is not considered systemic therapy.
* Diagnosed with immune deficiency or received systemic corticosteroid therapy or any other form of immunosuppressive therapy within 7 days before the first dose of investigational treatment. After consultation with the sponsor, the use of physiological doses of corticosteroids may be approved.
* Received liver radiotherapy within the past 2 weeks before enrollment.
* Known presence of central nervous system metastases and/or carcinomatous meningitis.
* Received systemic corticosteroid therapy within 7 days before enrollment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) | 1 year
  Time from initial drug administration to first radiographic disease progression or death (whichever occurs first).

SECONDARY OUTCOMES:
Overall response rate (ORR) | 1 year
  The proportion of subjects achieving complete response (CR) and partial response (PR) among the total subjects; includes assessment of both irradiated and non-irradiated lesions.
Disease control rate (DCR) | 1 year
  The proportion of subjects achieving complete response (CR), partial response (PR), and stable disease (SD) among the total subjects.
Overall survival (OS) | 3 year
  Time from initial drug administration to death of the subject for any reason.
The incidence and grade of adverse events | 2 year
  Common Terminology Criteria for Adverse Events (version 4.0) grades adverse event severity from 1=mild to 5=death.

CONTACTS AND LOCATIONS:
Overall Officials: Jin Bo Yue, Principal Investigator — Shandong Cancer Hospital and Institute
Locations (1):
- Jinbo Yue, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No